CLINICAL TRIAL: NCT06018467
Title: SENolytics to Improve Osteoporosis Therapy: a Randomised Controlled Clinical Trial The SENIOR Trial
Brief Title: Senolytics to Improve Osteoporosis Therapy
Acronym: SENIOR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EU CT: 2022-502076-23-00; 2022-502076-23-00 (Other: CTIS); NNF21OC0067839 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2023-08-23; First posted 2023-08-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Osteopenia, Osteoporosis; Age-related Bone Loss
Keywords: Age related bone loss; Cellular senescence; senolytic; senolytics; Dasatinib; Quercetin; NR; Nicoinamide riboside
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Dasatinib; Tablets; Quercetin; nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dasatinib plus Quercetin (DQ) (Experimental): Study participants will receive a combination of 100 mg/d dasatinib (oral) for two consecutive days and 1.250 mg/d quercetin (oral) for three consecutive days followed by 25 days without treatment, with treatment being repeated every 4 weeks for a total of 20 weeks (i.e., 5 times)
  Interventions: Drug: Dasatinib 100 Mg Oral Tablet; Dietary Supplement: Quercetin 1.250 mg (oral)
- Nicotinamide Riboside (NR) (Experimental): The participants will receive treatment with 1g Nicotinamide Riboside (oral) daily for 20 weeks
  Interventions: Dietary Supplement: Nicotinamide Riboside 1g (oral)
- Control (No Intervention): The participants in the Control group, will not receive any treatment for 20 weeks.

INTERVENTIONS:
Drug: Dasatinib 100 Mg Oral Tablet — Dasatinib tablets in blister packs of 10 tablets, from either: "Sandoz", "STADA Nordic", "Zentiva" or "Bristol-Myers Squibb"
  Other Names: Sprycel
  Arms: Dasatinib plus Quercetin (DQ)
Dietary Supplement: Quercetin 1.250 mg (oral) — five 200mg Quercetin Phytosome capsules, from Thorne
  Other Names: Quercetin Phytosome
  Arms: Dasatinib plus Quercetin (DQ)
Dietary Supplement: Nicotinamide Riboside 1g (oral) — four 250mg Nicotinamide Riboside Capsules, from Elysium Health
  Other Names: NR
  Arms: Nicotinamide Riboside (NR)

SUMMARY:
This randomised clinical trial aims to study osteoporosis as a disease of accelerated skeletal aging caused by the accumulation of senescent cells within the skeleton and investigate the effects and safety of senolytics and antioxidant therapy on bone.

DETAILED DESCRIPTION:
Background, hypothesis, and aim:

Evidence suggests that it is feasible to alleviate chronic age-related disorders by targeting the biology of aging. Recent studies implicate cellular senescence at the nexus of skeletal aging, suggesting that selectively eliminating senescent cells may emerge as a conceptually novel approach to manage the enormous problem of age-related bone loss. In addition, previous studies have demonstrated that antioxidants inhibit cellular senescence. The aim of this randomised clinical trial is to study osteoporosis as a disease of accelerated skeletal aging caused by accumulation of senescent cells within the skeleton and investigate the effects and safety of senolytics and antioxidant therapy on bone.

The main trial endpoint is the percent change in circulating marker of bone resorption (CTX) measured at baseline and at week 21. Secondary endpoints are the changes in bone resorption marker tartrate resistant acid phosphatase (TRAcP) and bone formation markers (PINP, osteocalcin, and bone alkaline phosphatase) measured at baseline and at 21 weeks.

Trial design:

The study design is a randomised controlled open-label clinical trial. Study participants will be randomised 1:1:1 to one of three treatment groups, that will include either,

1. a combination of 100 mg/d dasatinib (oral) for two consecutive days and 1.250 mg/d quercetin (oral) for three consecutive days followed by 25 days without treatment, with treatment being repeated every 4 weeks for a total of 20 weeks (i.e., 5 times), or
2. treatment with 1 g nicotinamide riboside (NR) (oral) daily for 20 weeks, or
3. no treatment for 20 weeks.

Each participant will have a total of 7 to 10 visits at the clinical site. Blood samples will be obtained at all but one visit (2x20 ml each time). ECG will be performed at 4-6 visits for group 1 and at 2 visits for group 2 and 3. Scans will be performed at the first two and the last visit. Muscle-function tests will be performed at 2nd and last visit. Bone biopsies for RNA-sequencing (a technique indicating which of the genes encoded in our DNA that are active) will be collected in those that provide a separate consent and in up to 20 participants in each group (using block randomisation to ensure balanced distribution of sex and age, equaling a maximum of 60 biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (menopause > 5 years and FSH and LH in the postmenopausal range) aged 60-90 years with increased fracture risk according to WHO 10 years absolute Fracture Risk Assessment Tool (FRAX)

  1. Osteopenia (ICD10 DM858A) based on a T-score ≤ -1 to -2.5 at the total hip/femoral neck, or lumbar spine, with or without a fragility fracture at any time (excluding hip and vertebral fractures within the last 2 years)
  2. osteoporosis (ICD10 DM819) based on a T-score between ≥-3 and ≤ -2.5, which includes candidates suitable for conventional osteoporosis therapies, but who prefer to participate in the trial, despite being candidates for conventional osteoporosis therapy, or candidates which cannot be treated with conventional therapies due to contraindications
* Ability to provide informed consent

Exclusion Criteria:

* DXA of hip or spine not possible e.g., due to a prosthesis
* Inability to provide fasting blood samples
* Primary hyperparathyroidism
* Vitamin D deficiency (<50 nM) (re-test after substitution acceptable)
* Known disorders affecting bone metabolism, e.g., uncontrolled thyrotoxicosis, chronic kidney disease defined as eGFR <30 or liver dysfunction, rheumatism, celiac disease/malabsorption, hypogonadism, severe COPD, hypopituitarism, Cushing's disease, uncontrolled diabetes (HbA1c > 58 mmol/mol).
* Antiresorptive or bone anabolic drugs for the last 2 years (5 years if treated with zoledronic acid)
* Concomitant treatments known to influence bone metabolism e.g., glucocorticoids (systemic treatments), anabolic steroids, etc.
* Subjects taking the following other drugs if they cannot be held for at least 2 days before and during administration of D+Q: digoxin, lithium, all statins, repaglidine, bosentan, gemfibrozil, olmesartan, enalapril, valsartan, methotrexate, corticosteroids, eluxadoline, eltrombopag, nitroglycerin, pioglitazone, glyburide, enzalutamide, ezetimibe, colchicine, imatinib, cyclosporine, tacrolimus, sirolimus, carbamazepine, flecainide, phenytoin, phenobarbital, rifampicin, theophylline, warfarin, heparin, clopidogrel, celecoxib, desipramine, thioridazine, venlafaxine, tizanidine, atomoxetine, voriconazole, citalopram, diazepam, escitalopram, propranolol, clozapine, cyclobenzaprine, mexiletine, olanzapine, ondansetron
* Subjects taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6 or strong inhibitors or inducers of CYP3A4 (e.g., cyclosporine, tacrolimus or sirolimus). If antifungals are necessary from an infectious disease perspective, then they will be allowed only if the levels are therapeutic.
* Subjects taking proton pump inhibitors and unwilling to discontinue therapy for two days before and during the study drug dosing periods.
* Anti-arrhythmic medications known to cause QTc prolongation
* Tyrosine kinase inhibitor therapy
* Subjects with an abnormal Complete Blood Count (clinically insignificant changes would be acceptable based on the judgement of the investigators)
* Subjects on antiplatelet agents (Clopidogrel; Dipyridamole + ASA; ASA, Ticagrelor; Prasugrel; Ticlopidine or other) who are unable or unwilling to reduce or hold therapy prior to and during the study drug dosing periods and collection of bone biopsies. Subjects may continue their previous regimen between study drug dosing periods.
* Known allergy to dasatinib, quercetin, or nicotinamide riboside
* Subjects taking the following antimicrobial agents: Aminoglycosides, Azole antifungals (fluconazole, miconazole, voriconazole, itraconazole), Macrolides (clarithromycin, erythromycin), antivirals (nelfinavir, indinavir, saquinavir, ritonavir, elbasvir/grazoprevir)
* Presence of any condition the Investigator believes would place the subject at risk or would preclude the subject from successfully completing all aspects of the trial e.g., heart failure, malignancy etc.
* QTc >470 msec
* Inability to take oral medication
* The study will exclude subjects with inability to speak and understand Danish and with inability to cooperate
* BMI ≥ 40

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Bone resorption marker CTX | Baseline, week 5, week 13, week 21
  Change in circulating marker of bone resorption C-terminal telopeptide of type I collagen (CTX) at 21 weeks.

SECONDARY OUTCOMES:
Bone resorption marker TRAcP | Baseline, week 5, week 13, week 21
  Change in circulating marker of bone resorption Tartrate Resistant Acid Phosphatase (TRAcP) at 21 weeks.
Bone formation markers (PINP, osteocalcin, and bone alkaline phosphatase) | Baseline, week 5, week 13, week 21
  Change in circulating markers of bone formation (PINP, osteocalcin, and bone alkaline phosphatase) at 21 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha Kassem, DMSc, PhD, Principal Investigator — Head of Research, Department of Endocrinology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
After completion of the project and irrespective of the outcomes, de-identified trial results will be published in peer-reviewed journals and www.clinicaltrials.gov. A summary of the clinical trial results will be presented in a language understandable to the layperson and made available in the EU database.